CLINICAL TRIAL: NCT06442228
Title: Investigation of the History of Polycystic Ovary Syndrome in First-degree Relatives of Male Partners of Couples Presenting for Infertility Treatment
Brief Title: History of Polycystic Ovary Syndrome in First-degree Relatives
Acronym: PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mujde Can Ibanoglu, Assoc. Prof, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024/05
Record Dates: First submitted 2024-05-14; First posted 2024-06-04 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: male; polycystic ovary syndrome; infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Individuals who have undergone spermiogram analysis at Etlik Zübeyde Hanım Gynecology Training and Research Hospital and whose first-degree relatives have a family history of PCOS will be included in the study group. Individuals who have undergone a spermiogram in our hospital, who fulfill the inclusion criteria and who do not have a family history of PCOS will be studied as a control group.
  Interventions: Diagnostic Test: spermiogram test

INTERVENTIONS:
Diagnostic Test: spermiogram test — Approximately 7 mL of blood sample will be taken by the health personnel in a vacuum gel tube for hormonal and biochemical analyses. The blood samples will be centrifuged at 1000xg for 20 minutes by the researchers. In the next step, the supernatant portion will be separated and transferred to 3 mL ependorfs. Serum samples will be stored in the -800C deep freezer of our hospital until the time of analysis.
  Sperm samples from individuals will be collected in our hospital in accordance with the protocol and the results will be reported.

SUMMARY:
The aim of this study was to investigate the semen analysis results of male patients with first-degree relatives meeting the diagnostic criteria for PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is an endocrine metabolic disorder characterised by menstrual irregularity, anovulation, clinical and/or biochemical signs of hyper androgenism (hirsutism and/or acne), micropolycystic ovaries and metabolic abnormalities.

This syndrome is clustered in family members and appears to be inherited through an oligogenic mechanism (1,2). As a result of familial clustering of the PCOS phenotype, metabolic risks have been shown to increase in family members, independent of gender.

The presence of a genetic background in the etiopathogenesis of PCOS means that men may also have signs and symptoms equivalent to PCOS. In addition, the genes responsible for PCOS susceptibility in women are also transferred to male relatives of these individuals. Hormonal and metabolic abnormalities have been identified in male relatives of women with PCOS. These men have shown a higher prevalence of early-onset (<35 years) androgenetic alopecia (AGA), type 2 DM and cardivascular diseases. In addition, prostate cancer, benign prostatic hyperplasia (BPH) and prostatitis have also been defined more frequently in this group of individuals (1,3).

In addition, differences in responses to gonadotropin-releasing hormone (GnRH) and FSH and LH levels were found in the brothers of women with PCOS compared to control groups.

According to genome studies (GWAS), FSHB gene on chromosome 11p14.1 represents the PCOS susceptibility focus in women (1). Genetic variations in FSHB affect male reproductive function. In fact, polymorphisms of the FSHB promoter have been associated with lower sperm count, higher LH, lower FSH and lower testicular volume (3,4).

In the light of this information, in this study, it was planned to evaluate the comparison of semen analysis results of male patients with a first-degree relative diagnosed with PCOS with the control group.

ELIGIBILITY:
Inclusion Criteria:

* The study will include male partners between the ages of 18-40 who have no known disease, who give spermiogram test for the evaluation of infertile couple in our hospital and who have accepted the consent form verbally and in writing.

Exclusion Criteria:

* Exclusion criteria;

  1. History of any chronic disease, urinary tract or reproductive disease, neurological or psychiatric condition in the male patient and recent fever (≥38°C in the last 3 months)
  2. Those with a history of vasectomy, cryptorchism, radiation history, chemotherapy, infections, sexual dysfunction and endocrine hypogonadism
  3. Especially those with a history of finasteride and dutasteride drug use.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
The results of male factors in male patients with first-degree female relatives who fulfill the diagnostic criteria for PCOS | 6 months
  sperm count

CONTACTS AND LOCATIONS:
Overall Officials: Yaprak Ustun, Study Director — Ankara Etlik Zubeyde Hanım Women's Health Training and Research Hospital, Ankara, Turkey.
Locations (1):
- Etlik Zübeyde Hanım, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Guardo F, Ciotta L, Monteleone M, Palumbo M. Male Equivalent Polycystic Ovarian Syndrome: Hormonal, Metabolic, and Clinical Aspects. Int J Fertil Steril. 2020 Jul;14(2):79-83. doi: 10.22074/ijfs.2020.6092. Epub 2020 Jul 15. PMID 32681618
- [Result] Cannarella R, Condorelli RA, Mongioi LM, La Vignera S, Calogero AE. Does a male polycystic ovarian syndrome equivalent exist? J Endocrinol Invest. 2018 Jan;41(1):49-57. doi: 10.1007/s40618-017-0728-5. Epub 2017 Jul 15. PMID 28711970
- [Result] Duskova M, Starka L. The existence of a male equivalent of the polycystic ovary syndrome--the present state of the issue. Prague Med Rep. 2006;107(1):17-25. PMID 16752800